CLINICAL TRIAL: NCT00108108
Title: An Open-label,Multi-center, Phase l/ll Study of Anti-CD40 Monoclonal Antibody (HCD122) Administered Intravenously to Subjects With Advanced Chronic Lymphocytic Leukemia That is Refractory or Relapsed After at Least One Previous Fludarabine-containing Chemotherapy Regimen
Brief Title: Dose-finding Trial of HCD122 in Patients With Chronic Lymphocytic Leukemia (CLL) That is Relapsed or Non-responsive to Prior Fludaribine Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment and minimal preliminary biological and clinical efficacy.
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHCD122A2101
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Lymphoid | interventions — lucatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HCD122 (Experimental)
  Interventions: Drug: HCD122

INTERVENTIONS:
Drug: HCD122

SUMMARY:
The purpose of this study is to determine the highest tolerated dose, safety and activity of HCD122 in patients with chronic lymphocytic leukemia who are relapsed after receiving prior treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CLL requiring treatment
* Refractory or relapsed disease
* Prior treatment with fludarabine
* Male or Female
* >18 years of age

Exclusion Criteria:

* Treatment with rituximab within 90 days and alemtuzumab or any monoclonal antibody within 6 months.
* Clinically significant cardiac dysfunction or other significant organ dysfunction

Additional eligibility criteria apply that will be reviewed with potential study subjects at the site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
to determine the maximum tolerated dose (MTD) | between study Day 1 and study Day 50

SECONDARY OUTCOMES:
to characterize safety and tolerability of HCD122 at each dose level in dose escalation patients | between study Day 1 and study termination
To characterize pharmacokinetics of HCD122 at each dose level in dose escalation patients | between study Day 1 and study termination
To characterize peripheral blood CD40 occupancy on CD5/CD19 (CLL) cells and CD5/CD19 cell depletion activity (pharmacodynamics) of HCD122 at each dose level in dose escalation patients | between study Day 1 and study termination
To assess preliminary anti-tumor activity of HCD122 in dose escalation patients | between study Day 1 and study termination

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Study Chair — Novartis
Locations (5):
- United States (5):
  - University of California San Diego StudyCoordinator:CHCD122A2101, La Jolla, California
  - St. Francis Cancer Research Foundation, Beech Grove, Indiana
  - The Sidney Kimmel Cancer Center at Johns Hopkins Hospital Div Of HematologicMalignancies, Baltimore, Maryland
  - OSU Medical Center/Arthur G. James Cancer Hospital StudyCoordinator:CHCD122A2101, Columbus, Ohio
  - MD Anderson Cancer Center/University of Texas Dept of MD Anderson CancerCent, Houston, Texas